CLINICAL TRIAL: NCT05467163
Title: CONDUCTion System Pacing Versus Biventricular Pacing After Atrioventricular Node Ablation in Heart Failure Patients With Symptomatic Atrial Fibrillation and Narrow QRS (CONDUCT-AF Trial)
Brief Title: Conduction System Pacing Versus Biventricular Pacing After Atrioventricular Node Ablation
Acronym: CONDUCT-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, David Žižek, MD, PhD, David Žižek, assist. prof., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONDUCT-AF trial
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Tachycardia-induced Cardiomyopathy; Atrial Fibrillation
Keywords: Heart failure; Atrial fibrillation; Conduction system pacing; His bundle pacing; Left bundle branch pacing; Biventricular pacing; Atrioventricular node ablation
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biventricular pacing + AV node ablation (Active Comparator): Implantation of biventricular pacemaker with or without defibrillator lead placement followed by AV node ablation. Optimal guidelines-based heart failure treatment.
  Interventions: Device: Biventricular pacemaker implantation; Procedure: AV node ablation
- Conduction system pacing + AV node ablation (Experimental): Implantation of permanent pacemaker with conduction system pacing (preferably left bundle branch) with or without defibrillator lead placement followed by AV node ablation. Optimal guidelines-based heart failure treatment.
  Interventions: Device: Conduction system pacing device implantation; Procedure: AV node ablation

INTERVENTIONS:
Device: Biventricular pacemaker implantation — Implantation of permanent pacemaker with biventricular stimulation with or without defibrillator lead placement using standard techniques. The right ventricle lead will be positioned in the RV apex or septum, while the left ventricle lead will be delivered to the most appropriate coronary sinus tributary, preferably posterolateral or lateral vein.
  Arms: Biventricular pacing + AV node ablation
Device: Conduction system pacing device implantation — Left bundle branch pacing (LBBP) will be the preferred pacing technique. In brief, after localizing the His bundle area the LBBP lead will be positioned approximately 1-1.5 cm distal to the His bundle position in the right ventricular septum. Before screwing the lead deep into the interventricular septum, the suitable position will be confirmed by fluoroscopic signs and adequate paced QSR morphology. Given that the pacing parameters with LBBP are typically low and stable, backup RV lead will not be mandatory. If LBBP will be unobtainable, His bundle pacing (HBP) implantation will be attempted. His bundle potential mapping will be performed with the use of the electrophysiological system and under fluoroscopic guidance. Distal HB potential with a large ventricular signal and a small atrial signal will be targeted before the pacing lead will be screwed into position. Backup RV lead will be mandatory for all patients receiving HBP devices.
  Arms: Conduction system pacing + AV node ablation
Procedure: AV node ablation — Atrioventricular node ablation (AVNA) will be performed following pacemaker implantation (preferably during the same hospitalization). After femoral vein access will be obtained, the ablation catheter will be positioned to the presumed area of the AV node in the mid-septum under fluoroscopy. The location will be optimized according to the intracardiac electrograms. Ablation will be performed in a temperature-controlled mode. Successful AVNA will be recognized with an abrupt drop of heart rate to 40 bpm and will continue for 60 seconds thereafter.

SUMMARY:
Atrioventricular node ablation (AVNA) with biventricular (BiV) pacemaker implantation is a feasible treatment option in patients with symptomatic refractory atrial fibrillation and heart failure. However, conduction system pacing (CSP) modalities, including His bundle pacing and left bundle branch pacing, could offer advantages over BiV pacing by providing more physiological activation. The randomized, interventional, multicentric study will explore whether CSP is non-inferior to BiV pacing in echocardiographic and clinical outcomes in heart failure (EF <50%) patients with symptomatic AF and narrow QRS scheduled for AVNA.

DETAILED DESCRIPTION:
Atrio-ventricular node ablation (AVNA) with subsequent permanent pacemaker implantation provides definite rate control and represents an alternative therapeutic approach in patients with symptomatic atrial fibrillation (AF) and rapid ventricular rate, refractory to optimal medical treatment or catheter ablation. However, optimal pacing modality remains unclear. Previous studies have demonstrated that biventricular (BiV) pacing followed by AVNA resulted in significant reduction in mortality, heart failure (HF) hospitalizations, significant improvement in symptoms and left ventricular (LV) remodeling. Although, its benefit was much less transparent in patients with narrow QRS and LV impairment, as it still causes abnormal cardiac activation with potential worsening of electrical dyssynchrony. To avoid the detrimental effects of BiV pacing a new concept, conduction system pacing (CSP), including His bundle Pacing (HBP) and left bundle branch pacing (LBBP), was proposed as a potential alternative. Both CSP modalities offer advantages over BiV pacing by providing more physiological activation, avoiding cardiac dyssynchrony and left ventricular dysfunction. Moreover, LBBP showed some advantages over HBP. Since the lead is implanted in the region of the left bundle, which has an adequate distance from the AVNA site, this modality could minimize the risk of increase in capture threshold after AVNA. Additionally, the pacing parameters of LBBP were stable in long-term follow-up studies precluding the need for back-up pacing. Therefore compared to HBP and BiV pacing, LBBP may offer a more feasible physiologic pacing option to be adopted into clinical practice. Some observational studies have already shown positive outcomes of HBP and LBBP in symptomatic AF patients who underwent AVNA with the favorable clinical and echocardiographic improvement compared to BIV pacing, especially in HF patients with narrow baseline QRS and reduced ejection fraction (EF<50%). However, prospective randomized study evaluating the value of CSP as an alternative approach to BiV pacing in combination with AVNA is lacking.

The purpose of this study is to compare the effects of CSP and conventional BiV pacing on echocardiographic and clinical outcomes in HF patients with symptomatic AF and narrow QRS scheduled for AVNA. In this multicentric study, 82 patients will be randomized into one of two arms: a BiV pacing arm with BiV pacemaker implantation + AVNA or CSP arm with the implantation of a CSP device + AVNA. In patients randomized in CSP group, LBBP will be the preferred pacing technique. If LBBP will be unobtainable, HBP implantation will be attempted. In both arms additional defibrillator backup will be implanted at the discretion of the physician according to the ESC guidelines. In short-term analysis after 6 months, echocardiographic, laboratory and symptomatic parameters will be evaluated. Long-term analysis to assess HF hospitalization, cardiovascular mortality and pacing parameters will be performed after at least 24 months of follow-up.

Investigators hypothesize that CSP could represent a feasible and safe alternative to BiV pacing in terms of clinical and echocardiographic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic permanent atrial fibrillation, refractory to drug therapy or failed catheter ablation
2. Left ventricular ejection fraction <50%
3. Narrow intrinsic QRS ≤ 120 ms
4. NT-proBNP > 600 ng/L
5. Patient has provided written informed consent
6. Age between 18 years and 85 years

Exclusion Criteria:

1. Pre-existing permanent pacemaker, implantable cardioverter-defibrillator or cardiac resynchronization device. Patients who had devices implanted that had <5% of paced beats (i.e., backup pacing) can be enrolled.
2. Life expectancy less than 12 months
3. Severe concomitant non-cardiac disease
4. Pregnancy
5. Recent (<3 months) myocardial infarction, percutaneous or surgical myocardial revascularization
6. Significant heart valve disease (severe insufficiency or stenosis)
7. Contraindication for oral anticoagulation
8. Mechanical tricuspid valve replacement
9. Unwillingness to participate or lack of availability for follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction. | baseline and 6 months
  Simpson's method assessed with echo.

SECONDARY OUTCOMES:
Time to the first occurrence of worsening heart failure or cardiovascular death. | at least 24 months
  An episode of heart failure that requires unplanned medical attention with increase of diuretic dose / intravenous diuretic therapy or death due to cardiovascular causes.
Time to the first occurrence of worsening heart failure. | at least 24 months
  An episode of heart failure that requires unplanned medical attention with increase of diuretic dose or intravenous diuretic therapy.
Time to cardiovascular death. | at least 24 months
  Death due to cardiovascular causes.
Number of heart failure hospitalizations. | at least 24 months
  Episodes of heart failure that require unplanned medical attention with increase of diuretic dose or intravenous diuretic therapy.
Change in LV end-diastolic and end-systolic volume index. | baseline and 6 months
  LV volumes indexed for body surface area - assessed by echo.
Change in clinical parameters | baseline and 6 months
  Quality of life measured by New York Heart Association (NYHA) classification.
Change in clinical parameters | baseline and 6 months
  Quality of life measured by Kansas City Cardiomyopathy Questionnaire (KCCQ).
Improvement in clinical parameters | baseline and 6 months
  Quality of life measured by European Heart Rhythm Association score of atrial fibrillation (EHRA AF).
Change in 6-Minute walk test. | baseline and 6 months
  Standard measurement.
Laboratory parameters. | baseline and 6 months
  NT-proB-type Natriuretic Peptide (BNP)
Procedural-related characteristics. | peri-procedural
  Total procedure and fluoroscopy time.
Procedure-associated adverse events. | peri-procedural, 30 days after the procedure
  Lead dislocations, device infection, bleeding, pneumotorax, etc.
Need for procedural reintervention. | at least 24 months
  Unplanned reintervention due to lead dysfunction or dislocation, device infection etc.
ECG parameters. | before and after the procedure
  QRS duration and morphology.
Pacing parameters. | peri-procedural, at least 24 months
  Capture threshold measurement.
Number of detected sustained VT/VF. | at least 24 months
  Detected sustained ventricular tachycardia or ventricular fibrillation on pacemaker telemetry.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Pernat, MD, PhD, Study Director — UMC Ljubljana; David Zizek, MD, PhD, Principal Investigator — UMC Ljubljana
Locations (10):
- University Hospital Graz - Divison of Cardiology, Graz, Austria
- Hospital Oost-Limburg (Hartzentrum Genk), Genk, Belgium
- Acibadem City Clinic Tokuda Hospital - Department of Invasive Electrophysiology, Sofia, Bulgaria
- Croatia (3):
  - Clinical Hospital Center Rijeka, Rijeka
  - University Hospital of Split, Split
  - University Hospital Centre Zagreb, Zagreb
- Central-Hospital of Northern Pest - Military Hospital, Budapest, Hungary
- County Clinical emergency hospital of Brasov - Department of Interventional Cardiology, Brasov, Romania
- Slovenia (2):
  - University Medical Centre Ljubljana - Department of cardiology, Ljubljana
  - University Medical Centre Ljubljana - Department of cardiovascular surgery, Ljubljana

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Tan ES, Rienstra M, Wiesfeld AC, Schoonderwoerd BA, Hobbel HH, Van Gelder IC. Long-term outcome of the atrioventricular node ablation and pacemaker implantation for symptomatic refractory atrial fibrillation. Europace. 2008 Apr;10(4):412-8. doi: 10.1093/europace/eun020. Epub 2008 Feb 12. PMID 18272509
- [Background] Orlov MV, Gardin JM, Slawsky M, Bess RL, Cohen G, Bailey W, Plumb V, Flathmann H, de Metz K. Biventricular pacing improves cardiac function and prevents further left atrial remodeling in patients with symptomatic atrial fibrillation after atrioventricular node ablation. Am Heart J. 2010 Feb;159(2):264-70. doi: 10.1016/j.ahj.2009.11.012. PMID 20152225
- [Background] Chatterjee NA, Upadhyay GA, Ellenbogen KA, Hayes DL, Singh JP. Atrioventricular nodal ablation in atrial fibrillation: a meta-analysis of biventricular vs. right ventricular pacing mode. Eur J Heart Fail. 2012 Jun;14(6):661-7. doi: 10.1093/eurjhf/hfs036. Epub 2012 Mar 21. PMID 22436544
- [Background] Brignole M, Pentimalli F, Palmisano P, Landolina M, Quartieri F, Occhetta E, Calo L, Mascia G, Mont L, Vernooy K, van Dijk V, Allaart C, Fauchier L, Gasparini M, Parati G, Soranna D, Rienstra M, Van Gelder IC; APAF-CRT Trial Investigators. AV junction ablation and cardiac resynchronization for patients with permanent atrial fibrillation and narrow QRS: the APAF-CRT mortality trial. Eur Heart J. 2021 Dec 7;42(46):4731-4739. doi: 10.1093/eurheartj/ehab569. PMID 34453840
- [Background] Muthumala A, Vijayaraman P. His-Purkinje conduction system pacing and atrioventricular node ablation. Herzschrittmacherther Elektrophysiol. 2020 Jun;31(2):117-123. doi: 10.1007/s00399-020-00679-7. Epub 2020 May 6. PMID 32377902
- [Background] Wang S, Wu S, Xu L, Xiao F, Whinnett ZI, Vijayaraman P, Su L, Huang W. Feasibility and Efficacy of His Bundle Pacing or Left Bundle Pacing Combined With Atrioventricular Node Ablation in Patients With Persistent Atrial Fibrillation and Implantable Cardioverter-Defibrillator Therapy. J Am Heart Assoc. 2019 Dec 17;8(24):e014253. doi: 10.1161/JAHA.119.014253. Epub 2019 Dec 13. PMID 31830874
- [Background] Su L, Cai M, Wu S, Wang S, Xu T, Vijayaraman P, Huang W. Long-term performance and risk factors analysis after permanent His-bundle pacing and atrioventricular node ablation in patients with atrial fibrillation and heart failure. Europace. 2020 Dec 26;22(Suppl_2):ii19-ii26. doi: 10.1093/europace/euaa306. PMID 33370800
- [Background] Huang W, Su L, Wu S, Xu L, Xiao F, Zhou X, Ellenbogen KA. Benefits of Permanent His Bundle Pacing Combined With Atrioventricular Node Ablation in Atrial Fibrillation Patients With Heart Failure With Both Preserved and Reduced Left Ventricular Ejection Fraction. J Am Heart Assoc. 2017 Apr 1;6(4):e005309. doi: 10.1161/JAHA.116.005309. PMID 28365568
- [Background] Zizek D, Antolic B, Meznar AZ, Zavrl-Dzananovic D, Jan M, Stublar J, Pernat A. Biventricular versus His bundle pacing after atrioventricular node ablation in heart failure patients with narrow QRS. Acta Cardiol. 2022 May;77(3):222-230. doi: 10.1080/00015385.2021.1903196. Epub 2021 Jun 2. PMID 34078244
- [Background] Ivanovski M, Mrak M, Meznar AZ, Zizek D. Biventricular versus Conduction System Pacing after Atrioventricular Node Ablation in Heart Failure Patients with Atrial Fibrillation. J Cardiovasc Dev Dis. 2022 Jul 1;9(7):209. doi: 10.3390/jcdd9070209. PMID 35877570
- [Background] Pillai A, Kolominsky J, Koneru JN, Kron J, Shepard RK, Kalahasty G, Huang W, Verma A, Ellenbogen KA. Atrioventricular junction ablation in patients with conduction system pacing leads: A comparison of His-bundle vs left bundle branch area pacing leads. Heart Rhythm. 2022 Jul;19(7):1116-1123. doi: 10.1016/j.hrthm.2022.03.1222. Epub 2022 Mar 26. PMID 35351624
- [Background] Brugada J, Katritsis DG, Arbelo E, Arribas F, Bax JJ, Blomstrom-Lundqvist C, Calkins H, Corrado D, Deftereos SG, Diller GP, Gomez-Doblas JJ, Gorenek B, Grace A, Ho SY, Kaski JC, Kuck KH, Lambiase PD, Sacher F, Sarquella-Brugada G, Suwalski P, Zaza A; ESC Scientific Document Group. 2019 ESC Guidelines for the management of patients with supraventricular tachycardiaThe Task Force for the management of patients with supraventricular tachycardia of the European Society of Cardiology (ESC). Eur Heart J. 2020 Feb 1;41(5):655-720. doi: 10.1093/eurheartj/ehz467. No abstract available. PMID 31504425